CLINICAL TRIAL: NCT01391065
Title: MR-PET Guided Biologically Optimised Interstitial Brachytherapy for Postoperative Recurrent Cervical Cancers
Brief Title: MR- PET Guided Biologically Optimised Interstitial Brachytherapy
Acronym: MR-PET Brachy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Associate Professor, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMH-IRB 843
Record Dates: First submitted 2011-07-01; First posted 2011-07-11 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Cervical Cancer
Keywords: Diffusion Weighted MRI; FLT PET; F-Miso PET; Image Guided Brachytherapy; Cervix; Postoperative Residual Disease/Postoperative recurrences
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): The study arm will undergo baseline multifunctional PET and MRI scans, before brachytherapy and at follow up
  Interventions: Radiation: MR PET Guided Brachytherapy

INTERVENTIONS:
Radiation: MR PET Guided Brachytherapy

SUMMARY:
The proposed two stage study will evaluate patterns of local recurrence after EBRT and brachytherapy in spatial reference to baseline functional MRI and FLT/F-Miso PET scan in patients undergoing chemoradiotherapy for postoperative recurrences of cervical cancer. The first stage of the study will focus on developing MR guided interstitial brachytherapy and validating the concept of high risk gross tumor volume (on the basis of functional imaging features).

The second stage thereafter will focus on developing biologically modulated interstitial brachytherapy.

In the proposed two staged study the investigators intend to prospectively evaluate and validate concept of HRGTV and develop technique of biologically dose modulated brachytherapy. The demonstration of technical feasibility and clinical safety of biologically modulated image guided radiotherapy in this pilot study for may pave the way for improving local control in patients with postoperative recurrences.

DETAILED DESCRIPTION:
Aims

Stage I

Aim 1: To spatially characterize biologically heterogenous subvolumes within the gross tumor through multimodality (18 F-Miso/FLT/Functional MR) image fusion.

Aim 2: To evaluate post external beam radiotherapy (EBRT) response in spatial reference to biological heterogeneous sub-volumes on imaging.

Stage II:

Aim 3: To evaluate technical feasibility of delivering dose modulated biologically optimized interstitial brachytherapy.

Aim 4: To evaluate acute and late toxicity and quality of life associated with biologically optimized brachytherapy

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* ECOG 0 or 1.
* Residual/ Recurrent tumor after hysterectomy of cervical cancer.
* No visceral metastasis.
* No known contraindication to contrast enhanced MRI/PET scan.
* Fit for radical treatment (radiotherapy+/-chemotherapy).

Exclusion Criteria:

* Expected survival less than 3 years due to coexisting morbid medical conditions precluding radical chemoradiotherapy.
* Inguinal or extra-pelvic nodal metastasis (Patients with common iliac nodal enlargement in the absence of paraaortic nodal metastasis on PET-CT may be included in the study).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02-23 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Local Response in spatial reference to High Risk GTV (as identified by functional imaging) | 3 months after treatment completion

SECONDARY OUTCOMES:
Incidence of Grade III rectal and bladder toxicity with biologically dose modulated brachytherapy | 2 years after treatment conclusion
  Stage II involves dose modulated brachytherapy wherein higher dose will be delivered to biologically high risk target volume. Saftey will be assessed initially by an interim analysis undertaken at 50 % accrual(median follow up 1 yr). If incidence of grade III-IV rectal and bladder toxicity >15% than the trial will be stopped else continued till target accrual. The technique will be considered to be safe if Grade III bladder and bowel toxicity remain to be under 15%.

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Centre of Treatment Research and Education In Cancer,Tata Memorial Centre, Navi Mumbai, Maharashtra, India

REFERENCES:
- [Derived] Chopra S, Engineer R, Shah S, Shukla R, Dora T, Gupta P, Paul SN, Popat P, Swamidas J, Mahantshetty U, Varghese L, Gupta S, Rangrajan V, Shrivastava S. MRI- and PET-Guided Interstitial Brachytherapy for Postsurgical Vaginal Recurrences of Cervical Cancer: Results of Phase II Study. Int J Radiat Oncol Biol Phys. 2020 Feb 1;106(2):310-319. doi: 10.1016/j.ijrobp.2019.10.037. Epub 2019 Nov 1. PMID 31682968
- Available data/document: Published article — https://doi.org/10.1016/j.ijrobp.2019.10.037